CLINICAL TRIAL: NCT05241067
Title: A Multicentric, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of Centhaquine as an Adjuvant to the Standard of Care in Patients With Moderate to Severe Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Multicentric, Randomized Study to Assess Safety and Efficacy of Centhaquine in Patients With ARDS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Centhaquine/ARDS /CT-2.2/2022
Record Dates: First submitted 2022-02-14; First posted 2022-02-15 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: ARDS; Resuscitation; Centhaquine; Hypoxia
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypoxia | interventions — Saline Solution; centhaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal saline (Placebo Comparator): Placebo (Dose: equal volume saline) + Standard of care
  Interventions: Drug: Normal Saline
- Centhaquine (Active Comparator): Centhaquine (Dose: 0.01 mg/kg) + Standard of care
  Interventions: Drug: Centhaquine

INTERVENTIONS:
Drug: Normal Saline — Placebo (Dose: equal volume saline) + Standard of care
  Other Names: Vehicle
  Arms: Normal saline
Drug: Centhaquine — Centhaquine (Dose: 0.01 mg/kg) + Standard of care
  Other Names: PMZ-2010
  Arms: Centhaquine

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a life-threatening condition with a diffuse, inflammatory form of lung injury, causing pulmonary infiltration and respiratory failure leading to poor oxygenation. It is a rapidly progressive form of respiratory failure and accounts for approximately 10% of admissions to the intensive care unit (ICU) and has a high mortality (40%) in severe cases. Globally, approximately 3 million ARDS cases are reported each year, with around 200,000 cases seen in the United States.

The etiology of ARDS could be pulmonary or extra-pulmonary. Patients with ARDS have symptoms like difficulty in breathing, shortness of breath, and cyanosis, and they may require assisted breathing/ventilatory support/extracorporeal membrane oxygenation. About 25% of ARDS patients need mechanical ventilation to support breathing; however, a ventilator-induced lung injury (VILI) is known to further exacerbate ARDS in many of them. In recent decades, numerous efforts have been made to develop therapies for treating/managing ARDS. Unfortunately, they have been largely unsuccessful or inconclusive, and at present, no effective pharmacological therapy for ARDS is available. Hence, development of better therapeutics for ARDS is an unmet need.

Centhaquine is a first-in-class resuscitative agent for hypovolemic shock approved for marketing in India. Centhaquine has been found to be an effective resuscitative agent in rat, rabbit, and swine models of hemorrhagic shock. Its safety and tolerability have been demonstrated in a human phase I study in 25 subjects (CTRI/2014/06/004647). Results from multicentric, randomized, double-blind, parallel, controlled clinical phase II (CTRI/2017/03/008184) and phase III (CTRI/2019/01/017196) studies conducted in India indicate that centhaquine is a novel, first-in-class, highly effective resuscitative agent for hypovolemic shock. A total of 155 patients with hypovolemic shock have been studied in the combined phase II and III trials, while a multicentric phase IV study (NCT05956418) in 400 patients with hypovolemic shock is currently being conducted in India. The outcomes of the completed trials indicate that centhaquine is safe and reduces mortality significantly (P=0.0271) compared to standard treatment of hypovolemic shock. In the phase II and III studies, ARDS and MODS were evaluated as secondary endpoints. Centhaquine provided hemodynamic stability and significantly reduced ARDS and multiple organ dysfunction score (MODS) in patients enrolled in these trials, which suggests that centhaquine has potential beyond treating hypovolemic shock and could be useful for ARDS treatment. Centhaquine is likely to provide hemodynamic stability, improve tissue oxygenation, reduce pulmonary edema, reduce ARDS score, and reduce MODS in patients with ARDS.

DETAILED DESCRIPTION:
This is a multicentric, randomized, double-blind, placebo-controlled phase-II clinical study to assess the safety and efficacy of centhaquine as an adjuvant to the standard of care in patients with moderate to severe ARDS. Approximately 10 study centers in the United States will participate in the study. For an individual patient, the duration of the study will be 60 days, including 3 study visits: visit 1/Day 1 (screening/randomization/baseline/treatment visit), visit 2/Day 28, and visit 3/End of Study (Day 60). At visit 1, approximately 80 eligible patients will be randomized 1:1 into 2 treatment groups of 40 each after meeting the eligibility criteria. A total of 40 patients will be enrolled in the centhaquine group (Group 1) and a total of 40 patients in the control group (Group 2):

* Group 1 (Active Group): Centhaquine (Dose: 0.01 mg/kg) + Standard of care
* Group 2 (Control group): Equal volume of Normal Saline + Standard of care In both treatment groups, patients will be provided with the standard of care. Centhaquine or Equal volume of Normal Saline will be administered intravenously after randomization to patients meeting the eligibility criteria. In the centhaquine group, centhaquine (0.01 mg/kg) dose will be administered as an intravenous (IV) infusion over 1 hour in 100 mL of normal saline. An additional dose of centhaquine will be administered on Day 2 if oxygenation and/or vasopressor support is required, but not before 24 hours of the previous dose (maximum 2 doses at an interval of 24 hours can be administered). In the control group, equal volume of normal saline will be administered as an intravenous (IV) infusion over 1 hour post-randomization. Conditions of administration will remain the same as for the centhaquine group. All subjects will be closely monitored during and after infusion. Vital signs will be monitored every 10 minutes during infusion. In the event of worsening hemodynamics or respiratory status, the infusion will be discontinued. Each subject will be monitored closely and followed up throughout his/her hospitalization. Moreover, he/she will be assessed for safety and efficacy parameters over 60 days from randomization.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in the study if he/she fulfills the following criteria:

1. Adult male or female aged 18 years or older
2. Hospitalized in the ICU diagnosed with moderate to severe ARDS having a PaO2/FiO2 ratio of < 200 mmHg or the SPO2/FiO2 ratio of ≤ 235( if SPO2 ≤ 97 %) with PEEP ≥ 5 cm H20 include the patient receiving invasive /non-invasive ventilation (NIV/CPAP).
3. The first dose of the study drug should be administered within 48 hours of confirming moderate to severe ARDS.
4. Requires vasopressor support
5. Written informed consent

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if he/she meets any of the following exclusion criteria:

1. Receiving or expected to receive extracorporeal membrane oxygenation or high-frequency oscillatory ventilation
2. Confirmed pregnancy
3. Breast feeding
4. Participating in another interventional study
5. Requires or having the renal replacement therapy
6. Hepatic failure (Child-Pugh scores B and C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of PaO2/FiO2 ratio ≥200 mmHg or relative increase by 50 mmHg from baseline | 3 days
  The study's primary objective is to determine the clinical effect of centhaquine in patients with moderate to severe ARDS.

SECONDARY OUTCOMES:
28-day all-cause mortality | 28 days
  Incidence of 28-day all-cause mortality
60-day all-cause mortality | 60 days
  Incidence of 60-day all-cause mortality
Time to clinical improvement on WHO 8-point ordinal scale | 60 days
  Time to clinical improvement on WHO 8-point ordinal scale (ranging from 1-Ambulatory to 8-Death)
Hospital free days | 28 days
  Hospital free days [Time frame: The number of days beginning with the day of randomization counted as "Day 1" through Day 28]
ICU free days | 28 days
  • ICU free days [Time frame: The number of days beginning with the day of randomization counted as "Day 1" through Day 28]
Ventilator free days (VFDs) | 28 days
  Ventilator free days (VFDs) in hospital [Time frame: The number of days beginning with the day of the episode counted as "Day 1 through Day 28, during which the patient is being cared for in the hospital]
Days alive free of renal replacement therapy | 28 days
  • Days alive free of renal replacement therapy [Time frame: The number of days beginning with the day of randomization counted as "Day 1" through Day 28]
Days alive free of vasopressor(s) | 28 days
  Days alive free of vasopressor(s) [Time frame: The number of days beginning with the day of randomization counted as "Day 1" through Day 28]
A ≥ 50% reduction in vasopressor(s) (norepinephrine equivalents; NEE) dose. | 3 days
  The proportion of patients who have a ≥ 50% reduction of vasopressor(s) (norepinephrine equivalent; NEE) dose from the time of randomization [Time frame: 24 hours, 48 hours, 72 hours from the time of randomization].
Change in blood lactate | 3 days
  Change in blood lactate [Time frame: Day 1 through Day 3]
Change in Sequential Organ Failure Assessment (SOFA) Score | 9 days
  • Change in Sequential Organ Failure Assessment (SOFA) score [Time frame: baseline through Day 9 or at the time of hospital discharge, whichever is earlier.]
Adverse events (AEs) and serious adverse events (SAEs) | 28 days
  Proportion of patients with adverse events (AEs) and serious adverse events (SAEs)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulati A, Choudhuri R, Gupta A, Singh S, Ali SKN, Sidhu GK, Haque PD, Rahate P, Bothra AR, Singh GP, Maheshwari S, Jeswani D, Haveri S, Agarwal A, Agrawal NR. A Multicentric, Randomized, Controlled Phase III Study of Centhaquine (Lyfaquin(R)) as a Resuscitative Agent in Hypovolemic Shock Patients. Drugs. 2021 Jun;81(9):1079-1100. doi: 10.1007/s40265-021-01547-5. Epub 2021 Jun 1. PMID 34061314
- [Background] Ranjan AK, Zhang Z, Briyal S, Gulati A. Centhaquine Restores Renal Blood Flow and Protects Tissue Damage After Hemorrhagic Shock and Renal Ischemia. Front Pharmacol. 2021 May 3;12:616253. doi: 10.3389/fphar.2021.616253. eCollection 2021. PMID 34012389
- [Background] Gulati A, Jain D, Agrawal NR, Rahate P, Choudhuri R, Das S, Dhibar DP, Prabhu M, Haveri S, Agarwal R, Lavhale MS. Resuscitative Effect of Centhaquine (Lyfaquin(R)) in Hypovolemic Shock Patients: A Randomized, Multicentric, Controlled Trial. Adv Ther. 2021 Jun;38(6):3223-3265. doi: 10.1007/s12325-021-01760-4. Epub 2021 May 10. PMID 33970455
- [Background] Kontouli Z, Staikou C, Iacovidou N, Mamais I, Kouskouni E, Papalois A, Papapanagiotou P, Gulati A, Chalkias A, Xanthos T. Resuscitation with centhaquin and 6% hydroxyethyl starch 130/0.4 improves survival in a swine model of hemorrhagic shock: a randomized experimental study. Eur J Trauma Emerg Surg. 2019 Dec;45(6):1077-1085. doi: 10.1007/s00068-018-0980-1. Epub 2018 Jul 13. PMID 30006694
- [Background] Briyal S, Gandhakwala R, Khan M, Lavhale MS, Gulati A. Alterations in endothelin receptors following hemorrhage and resuscitation by centhaquin. Physiol Res. 2018 Jun 27;67(Suppl 1):S199-S214. doi: 10.33549/physiolres.933856. PMID 29947540
- [Background] Papalexopoulou K, Chalkias A, Pliatsika P, Papalois A, Papapanagiotou P, Papadopoulos G, Arnaoutoglou E, Petrou A, Gulati A, Xanthos T. Centhaquin Effects in a Swine Model of Ventricular Fibrillation: Centhaquin and Cardiac Arrest. Heart Lung Circ. 2017 Aug;26(8):856-863. doi: 10.1016/j.hlc.2016.11.008. Epub 2016 Dec 19. PMID 28385449
- [Background] O'Donnell JN, O'Donnell EP, Kumar EJ, Lavhale MS, Andurkar SV, Gulati A, Scheetz MH. Pharmacokinetics of centhaquin citrate in a dog model. J Pharm Pharmacol. 2016 Jun;68(6):803-9. doi: 10.1111/jphp.12554. Epub 2016 Apr 25. PMID 27109141
- [Background] O'Donnell JN, Gulati A, Lavhale MS, Sharma SS, Patel AJ, Rhodes NJ, Scheetz MH. Pharmacokinetics of centhaquin citrate in a rat model. J Pharm Pharmacol. 2016 Jan;68(1):56-62. doi: 10.1111/jphp.12498. Epub 2016 Jan 4. PMID 26725913
- [Background] Papapanagiotou P, Xanthos T, Gulati A, Chalkias A, Papalois A, Kontouli Z, Alegakis A, Iacovidou N. Centhaquin improves survival in a swine model of hemorrhagic shock. J Surg Res. 2016 Jan;200(1):227-35. doi: 10.1016/j.jss.2015.06.056. Epub 2015 Jun 29. PMID 26216751
- [Background] Gulati A, Zhang Z, Murphy A, Lavhale MS. Efficacy of centhaquin as a small volume resuscitative agent in severely hemorrhaged rats. Am J Emerg Med. 2013 Sep;31(9):1315-21. doi: 10.1016/j.ajem.2013.05.032. Epub 2013 Jul 19. PMID 23871440
- [Background] Lavhale MS, Havalad S, Gulati A. Resuscitative effect of centhaquin after hemorrhagic shock in rats. J Surg Res. 2013 Jan;179(1):115-24. doi: 10.1016/j.jss.2012.08.042. Epub 2012 Sep 2. PMID 22964270
- [Background] Gulati A, Lavhale MS, Garcia DJ, Havalad S. Centhaquin improves resuscitative effect of hypertonic saline in hemorrhaged rats. J Surg Res. 2012 Nov;178(1):415-23. doi: 10.1016/j.jss.2012.02.005. Epub 2012 Apr 2. PMID 22487389